CLINICAL TRIAL: NCT03452904
Title: The Randomized FADDY Study (FrActional Flow Reserve Guided Drug Coated Balloon Only Strategy in De Novo coronarY Lesions)
Brief Title: FrActional Flow Reserve Guided Drug Coated Balloon Only Strategy in De Novo coronarY Lesions (FADDY)
Acronym: FADDY
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHZJU CT008
Record Dates: First submitted 2018-02-22; First posted 2018-03-02 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2017-12

CONDITIONS: Coronary Stenosis
Keywords: In suit coronary lesions; Drug-coated balloon; Drug-eluting stent; Restenosis
MeSH Terms: conditions — Coronary Stenosis | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug-coated balloon (Experimental): Treatment of in suit coronary lesions with drug-coated balloon
  Interventions: Device: Drug-coated balloon
- Drug-eluting stent (Active Comparator): Treatment of in suit coronary lesions with drug-eluting stent
  Interventions: Device: Drug-eluting stent

INTERVENTIONS:
Device: Drug-coated balloon — Treatment of in suit coronary lesions with drug-coated balloon
  Arms: Drug-coated balloon
Device: Drug-eluting stent — Treatment of in suit coronary lesions with drug-eluting balloon
  Arms: Drug-eluting stent

SUMMARY:
Drug-eluting stent (DES) has been the primary choice for in suit coronary lesions treatment. In comparison to bare-metal stent (BMS), it evidently decreases the rate of restenosis. However, in recent years in-stent restenosis or thrombogenesis caused by acquired stent malapposition in the late stage or by new in-stent atherosclerotic plaques was oberved, which possibly was associated with chronic inflammation stimulation because of residual intravascular metal or polymer coating. Through being expanded around 30 to 60 seconds, drug-coated balloon (DCB) can ensure adequate paclitaxel enter the artery wall, which can inhibit smooth muscle cells hyperplasia without remaining any foreign body. In recent small sample trials, they showed that sole DCB treatment had a good long-term effect when pre-treating ideal in suit coronary lesions (defined as residual stenosis< 30%, without dissection severer than type C, anterograde flow TIMI III). In PEPCAD I trial, the rate of major adverse cardiovascular events (MACE) was 6.1% in the first 12 months and persistent to 3-year follow up. Small sample prospective observational study from Korea, like Shin, showed that in the in suit coronary lesions with the fractional flow reserve (FFR)>0.85 after percutaneous transluminal coronary angioplasty (PTCA), the FFR kept unchanged in the 9-month follow up after DCB treatment and there was not MACE happened. However, so far randomized controlled trials with large sample to confirm their non-inferiority compared with DES when treating relatively larger in suit coronary lesions are lacked. Meanwhile, a number of doctors worried about acute cardiovascular occlusion and long-term restenosis. In this study, we assume that in the in suit coronary lesions with FFR>0.85 after PTCA pre-treatment, DCB treatment is not inferior to DES treatment regarding to middle- and long-term functional recovery.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Criteria:

  1. Patients with age >= 18 years old
  2. Patients with coronary artery disease is confirmed by angiography
  3. Patients with angina (CCS class II-IV) or documented ischemia evidence with ECG or ECT
  4. Patients agree to sign the informed consent
* Angiographic Criteria:

  1. In suit coronary lesions
  2. Reference diameters of target vessels by visual estimation from 2.5 mm to 3.5 mm and < 28 mm in length
  3. Lesion diameter stenosis >= 70% by visual estimation or >= 50% with objective ischemia evidence (exercise stress testing, ECT or FFR< 0.8)

Exclusion Criteria:

* Clinical Criteria:

  1. Patients with STEMI <= 1 week
  2. Patients with LVEF < 30%
  3. Patients with bleeding diathesis or known anticoagulation dysfunction
  4. Patients with medical history regarding of intracranial tumor, aneurysm, arteriovenous malformation or cerebral apoplexy; stroke or TIA within 6 months; gastrointestinal hemorrhage within 2 months; major surgery within 6 weeks; recent or known platelet < 100,000/mm3 or hemoglobin < 10 g/dL
  5. Patients with planed selective operation probably leading to stopping using ADP receptor antagonists in advance
  6. Patients with life expectancy is less than 1 year because of combined comorbidity of other system
* Angiographic Criteria:

  1. Acute thrombotic lesions
  2. Left main coronary artery lesions
  3. Severe intima tear lesions
  4. Coronary artery bypass grafts lesions
  5. In-stent restenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
9-month fractional flow reserve value | 9 months

SECONDARY OUTCOMES:
Late lumen loss | 9 months
Percent restenosis | 9 months
Failure rate of target lesions | 9 months
Rate of thrombosis in target lesions | 9 months
Cumulative MACE rate | 9 months
Success rate of the strategy | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Jian-an Wang, MD,PhD, Study Chair — Second Affiliated Hospital of Zhejiang University, School of Medicine
Locations (1):
- Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China